CLINICAL TRIAL: NCT02106026
Title: Effectiveness of a Nursing Education Intervention on Duration of Breastfeeding and on Post-natal Breast Complications in Primiparous Women: a Randomized Controlled Trial
Brief Title: Nursing Education Intervention for Maternal Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Concepcion Carratala-Munuera, Dr, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LACT-120413
Record Dates: First submitted 2014-03-28; First posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Breast Feeding; Postpartum Breast Disorders
Keywords: Breastfeeding; Nursing; Patient Education as Topic; Health Knowledge, Attitudes, Practice; Hispanic Americans.
MeSH Terms: conditions — Breast Feeding; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional (No Intervention): All expectant mothers received the usual information about the advantages of maternal milk during pre-natal period. Nurses provided the information in personalized dialogue with the women during obstetric consultations.
- Preventive education (Experimental): It was provided by the nurses during obstetric consultation in pre-natal period and averaged 30 minutes in duration. The intervention group received education to facilitate successful breastfeeding and symptom management as nipple pain. This was supported by strategies designed to (1) prevent problems associated with breastfeeding (nipple lesions, cracks and mastitis), (2) perform breast-care procedures, (3) strengthen information about the advantages of maternal breastfeeding (nutritional support, importance as food for the baby, availability, post-partum recovery) and (4) provide asepsis and hygiene measures. The nurses encouraged participation and gave the education in personalized dialogue with the woman. The information was reinforced with an illustrated explanatory leaflet.
  Interventions: Other: Preventive education

INTERVENTIONS:
Other: Preventive education — The intervention group received education to facilitate successful breastfeeding and symptom management as nipple pain. This was supported by strategies designed to (1) prevent problems associated with breastfeeding (nipple lesions, cracks and mastitis), (2) perform breast-care procedures, (3) strengthen information about the advantages of maternal breastfeeding (nutritional support, importance as food for the baby, availability, post-partum recovery) and (4) provide asepsis and hygiene measures.
  Arms: Preventive education

SUMMARY:
An antenatal education intervention in primiparous women improves breastfeeding duration and reduces post-natal complications.

DETAILED DESCRIPTION:
A randomized controlled clinical trial of an educational intervention was undertaken at a public hospital. the investigators compared a health education based on techniques to prevent complications and increase information about the benefits of breastfeeding with the usual practice. A group of nurses delivered the educational intervention. The trial involved randomization of 314 primiparous women. The analysis was by 'intention-to-treat'.

ELIGIBILITY:
Inclusion Criteria:

* primiparous women,
* no contraindications to breastfeeding,
* no skin disorders,
* no breast surgery,
* voluntary provision of data to enable their later localization.

Exclusion Criteria:

* women who planned to deliver their babies in other hospitals,
* twin pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2004-12; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Breastfeeding duration | At 6 months postpartum
Breastfeeding duration | At 1 month postpartum

SECONDARY OUTCOMES:
Knowledge about breastfeeding and care of the breasts, | Inmediate postpartum period.
Incidence of mothers with post-natal breast complications, such as cracks, breast lesions or mastitis | At 1 month postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Concepcion Carratala-Munuera, PhD, Principal Investigator — Universidad Miguel Hernandez de Elche